CLINICAL TRIAL: NCT00609089
Title: A Stage 1 Study of Community Reinforcement and Family Training for Treatment Drug Abuse Treatment Retention/HIV Risk Reduction
Brief Title: Community Reinforcement and Family Training for Drug Abuse Treatment Retention/HIV Risk Reduction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Maryhaven (Unknown)
Responsible Party: Principal Investigator, Gregory S. Brigham, Clin Research Admin/Dir, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5K23DA021512-02 (NIH); 5K23DA021512-02 (NIH)
Record Dates: First submitted 2008-01-22; First posted 2008-02-06 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Heroin Dependence; Opiate Dependence; Substance Dependence
Keywords: Family; treatment; reinforcement; substance; trial; drug; abuse; HIV; risk
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Community Reinforcement and Family Training for Retention in Treatment and Recovery and Reduction of HIV Risk Behavior (CRAFT-T)
  Interventions: Behavioral: CRAFT-T
- II (Active Comparator): Treatment As Usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: CRAFT-T — The Community Reinforcement and Family Training for Treatment Retention and HIV Risk Reduction treatment (CRAFT-T) was be developed in phase 1 and 2 of the current study and consists of twelve manual-guided weekly one-hour individual sessions for the concerned significant other and 2 one hour sessions for the identified patient. The intervention also allows for up to two additional sessions (total of 14 visits) to help arrange re-entry into substance abuse treatment when needed. The identified patient receives this intervention in addition to the usual services at the drug treatment program (Maryhaven).
  Arms: I
Behavioral: Treatment as usual — Treatment as usual will be the normal course of treatment for concerned significant others (CSOs) in the outpatient department.
  Arms: II

SUMMARY:
The planned research will adapt an intervention of known efficacy to target a new outcome of significant importance to public health. Specifically the Community Reinforcement and Family Training (CRAFT) procedures will be adapted, from reinforcing treatment entry, to reinforcing treatment retention and HIV risk behavior reduction in persons with opioid dependence who receive a Buprenorphine taper detoxification. The research plan includes three phases: 1) development of a manual guided therapy, 2) development of therapist training and fidelity measures and 3) a randomized pilot evaluation with 52 patients receiving either the new CRAFT treatment or treatment as usual.

ELIGIBILITY:
Concerned Significant Other Inclusion Criteria: 1)be a first-degree relative, spouse, or intimate partner, or plan to live with the IP following the IP's detoxification, must plan to have contact with the IP at least 40% of the first 90 days post randomization, 2)be age 18 or older, 3)live within approximately 60 miles of Maryhaven, )be willing to participate in the protocol (i.e., to be randomized to treatment, to attend regular treatment sessions, to have their sessions audio taped, etc.), 5)be willing to sign a HIPAA-compliant release(s) of information to allow research staff access to any information collected from this subject during the study. Such staff may include RAs, therapists, supervisors, data managers, statisticians, QA personnel, etc., 6)be able to understand and provide written informed consent in English, 7)express desire to assist the IP with treatment retention and HIV risk behavior reduction.

Concerned Significant Other Exclusion Criteria: 1) are unlikely to be available to complete the entire protocol (e.g., plan to relocate, intention to not continue if assigned to a perceived unattractive arm of the study), 2)have a condition (e.g., medical complications, psychiatric problems, etc.) that would necessitate inpatient treatment or would make study participation difficult, 3)have engaged in domestic violence or assault within the previous year or have a history of severe violence (i.e., use of a weapon or violence leading to a hospitalization). For the purposes of the present protocol, domestic violence is defined as any physical abuse between intimately involved partners, roommates, or family members, 4)are currently at risk for suicide as evidenced by presence of at least one of the following; a) a history of a suicide attempt(s) and current suicidal ideation, b) current suicide ideation including recurrent thoughts of suicide with intention to harm themselves, c) persistent or recurring desire to die, d) a plan to harm themselves, e) indication that they would not take steps to save their own life, 5)have been the victim of severe domestic violence (i.e., use of a weapon or violence leading to a hospitalization) by the IP.

Identified Patient Inclusion Criteria: 1)be a first-degree relative, spouse, or intimate partner of the CSO, or someone who lives with the CSO, 2)be age 18 or older, 3)be currently enrolled in the BUP/NX 13-day taper protocol in Maryhaven's detoxification program, 4)intend to continue with outpatient treatment at Maryhaven, 5)be willing to participate in the protocol (i.e., to be randomized to treatment, to attend regular treatment sessions, to have their sessions audio taped, etc.), 6)be willing to sign a HIPAA compliant release(s) of information to allow research staff access to any information collected from this subject during the study. Such staff may include RAs, therapists, supervisors, data managers, statisticians, QA personnel, etc., 7)be able to understand and provide written informed consent in English, and 8)have a substance use disorder assessed by the Structured Clinical Interview for DSM-IV.

Identified Patient Exclusion Criteria: 1)have engaged in domestic violence or assault within the previous year or have a history of severe violence (i.e., use of a weapon or violence leading to a hospitalization), 2)have a history of a suicide attempt(s)within the past year or current suicidal ideation, 3)are currently at risk for suicide as evidenced by presence of at least one of the following; (same as CSO suicide lethality criteria above), 4)have a condition (e.g., medical complications, or psychiatric problems other than substance abuse, etc.) that would necessitate residential/inpatient treatment or would make study participation difficult, 5)under a court order to enter and remain in treatment program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is retention in drug abuse treatment, specifically time to first drop from services for at least 3 weeks duration. | 6 months

SECONDARY OUTCOMES:
The Identified Patient's engagement in behaviors that increase the risk of contracting HIV, as measured by the RAB | 6 months
The concerned significant other's (CSO's) engagement in behaviors that increase the risk of contracting HIV, as measured by the RAB, | 6 months
The identified patient's successful completion of drug abuse treatment episode | 6 months
The portion of available treatment sessions attended during each assessment period including, | 6 months
Substance use (defined as days of self-reported substance use, with partial confirmation by urinalysis and breathalyzer) during the active study phase and through the 3 month and 6-month follow-ups. | 6 months
The identified patient's substance use as reported by the CSO (collateral reports of drug use). | 6 months
Changes in concerned significant other and identified patient function as measured using the Brief Symptom Inventory. Specifically, the Global Severity Index (GSI) score. | 6 months
Concerned significant other and identified patient's relationship satisfaction (the score on the General Happiness Scale of the RHS). | 6 months
Marital satisfaction as measured by the KMS for the sub-sample of concerned significant others who are married to their identified patient's. | 6 months
The identified patient's (IP) retention in any substance abuse specific intervention, including self-help, as reported by the IP on the Treatment tracking form. | 6 months
The identified patient's retention in any substance abuse specific intervention, including self-help, as reported by CSO on the Treatment Tracking form. | 6 months
Identified patient (IP) attendance at self-help groups (i.e., AA, NA, CA) (defined as the number of times that the IP has attended a self-help group as assessed on the Treatment Services Review). | 6 months
Identified patient's use of professional services, other than substance abuse treatment, as reported on the TSR. | 6 months
Concerned significant others satisfaction with treatment as measured by the Participant Satisfaction Form. | 3 months
Identified patient's satisfaction with treatment as measured by the Participant Satisfaction | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Gregory S. Brigham, Ph.D., Principal Investigator — University of Cincinnati
Locations (1):
- Maryhaven, Columbus, Ohio, United States

REFERENCES:
- [Background] Garner BR, Barnes B, Godley SH. MONITORING FIDELITY IN THE ADOLESCENT COMMUNITY REINFORCEMENT APPROACH (A-CRA): THE TRAINING PROCESS FOR A-CRA RATERS. J Behav Anal Health Sports Fit Med. 2009 Spring;2(1):43-54. doi: 10.1037/h0100373. PMID 21533009